CLINICAL TRIAL: NCT04980989
Title: A Prospective Randomized Trial of Interactive Telemonitoring in the Follow-up of Patients Treated for Breast Cancer
Brief Title: Follow-up of Early Breast Cancer (BC) Patients by Telephone or Mobile Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other); Noona Healthcare (Unknown)
Responsible Party: Principal Investigator, Johanna Mattson, Physician-in-Chief, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 112/13/03/02/2015
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer, Early-Onset
Keywords: follow-up, mobile software, early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with early breast cancer were randomized at the final visit of adjuvant radiotherapy to surveillance by phone calls or by mobile Noona software. After six months the groups were crossed over to the other arm. At 12 months the patients were asked their preference. At baseline, 6 months and 12 months the patients answered the other questionnaires on patient satisfaction, quality of life, symptoms and use of other healthcare services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile software (Experimental): Patient with early breast cancer were followed-up by mobile software for the first six months. At six months they crossed-over to be followed-up by telephone calls for the next six months.
  Interventions: Device: Mobile software for follow-up of early breast cancer
- Telephone calls (Active Comparator): Patient with early breast cancer were followed-up by telephone calls for the first six months. At six months they crossed-over to be followed-up by mobile software for the next six months.
  Interventions: Device: Mobile software for follow-up of early breast cancer

INTERVENTIONS:
Device: Mobile software for follow-up of early breast cancer — The patients were randomized to use mobile software or telephone calls as the follow-up modality for early breast cancer
  Other Names: Noona mobile software

SUMMARY:
Patients with early breast cancer were randomized at the final visit of adjuvant radiotherapy to surveillance by phone calls or by mobile Noona software. After six months the groups were crossed over to the other arm. At 12 months the patients were asked their preference which was the primary end-point. At baseline, 6 months and 12 months the patients answered the other questionnaires.

DETAILED DESCRIPTION:
Patients with early breast cancer were randomized at the final visit of adjuvant radiotherapy to surveillance by phone calls or by mobile Noona software. After six months the groups were crossed over to the other arm.

The primary end point was to find out patient preference for the modality of surveillance. Secondary endpoints were patient satisfaction, symptoms, quality of life and cost of follow-up during surveillance modalities.

At 12 months the patients were asked their preference for the follow-up modality of early breast cancer. At baseline, 6 months and 12 months the patients answered the other questionnaires on quality of life, symptoms, patient satisfaction and use of other health-care services. Information on the cost of follow-up was gathered from the hospital and other registries.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with early breast cancer after primary treatment including also radiotherapy (the patients were randomized at the final visit of radiotherapy)

Exclusion Criteria:

* not able to use a computer
* another malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 765 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Patient preference for follow-up modality | At 12 months during follow-up of early breast cancer
  Questionnaire of patient preference

SECONDARY OUTCOMES:
Quality of life during follow-up modality | At baseline, 6 months and 12 months
  Quality of life questionnaires
Patient satisfaction | At 6 months and 12 months
  Patient satisfaction questionnaires
Symptoms | At baseline, 6 months and 12 months
  Symptom questionnaire
Use of other healthcare services | At 6 months and 12 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Mattson, MD, PhD, Principal Investigator — Helsinki University Central Hospital; Carl Blomqvist, Professor, Study Chair — Helsinki University Central Hospital; Johanna Mattson, MD, PhD, Study Director — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mattson J, Peltola M, Poikonen-Saksela P, Hermanson T, Their J, Farkkila N, Roine R, Blomqvist C. Digital solution in the follow-up of early breast cancer a randomized study. Acta Oncol. 2023 May;62(5):513-521. doi: 10.1080/0284186X.2023.2212409. Epub 2023 May 16. PMID 37190970